CLINICAL TRIAL: NCT00890591
Title: National, Multicenter, Open-Label and Prospective Study Assessment of Efficacy and Safety in Stage 1 and 2 Essential Hypertension With Olmesartan Medoxomil Based Treatment Algorithm From Monotherapy to Association With Hydrochlorothiazide and Amlodipine Besylate
Brief Title: Efficacy and Safety of Olmesartan Medoxomil in Stage 1 and 2 Essential Hypertension
Acronym: Benibest
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Medical Affairs Manager, Daiichi Sankyo Brazil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPB-OM-0106
Record Dates: First submitted 2009-02-11; First posted 2009-04-30 (Estimated); Results first posted 2009-04-30 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-05

CONDITIONS: Essential Hypertension
Keywords: hypertension; angiotensin II type 1 receptor blocker; olmesartan
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — Olmesartan Medoxomil; Hydrochlorothiazide; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: olmesartan medoxomil + hydrochlorothiazide, if necessary + amlodipine, if necessary

INTERVENTIONS:
Drug: olmesartan medoxomil + hydrochlorothiazide, if necessary + amlodipine, if necessary — olmesartan medoxomil tablets,or olmesartan medoxomil/hydrochlorothiazide tablets, if necessary + amlodipine tablets, if necessary. All interventions are once-daily for 4 to 9 weeks

SUMMARY:
In patients naive to treatment or after a 2-week washout period for patients whose treatment was ineffective, the use of olmesartan was assessed in a 4-phase treatment scheme: monotherapy, addition of hydrochlorothiazide (2 phases), addition of amlodipine.

ELIGIBILITY:
Inclusion Criteria:

* Stage 1 and 2 hypertension without treatment for at least 2 weeks
* Women with no risk of becoming pregnant

Exclusion Criteria:

* Study participation could result in risk to health of subject
* Cardiovascular disease
* Secondary hypertension or stage 3 hypertension
* Myocardial infarction within the last 6 months
* Congestive heart failure
* Pulmonary edema
* Valvular alterations or rheumatic cardiopathy
* Clinically relevant conduction disorders significant arrhythmias
* Alcohol or illicit drug use
* Medication abuse
* Pregnant or nursing women

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2006-08; Primary Completion 2007-06 (Actual); Study Completion 2007-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study pop. was defined by the inclusion criteria. This study was carried out in 14 centers in Brazil with inclusion 2 months after the first study subject, started in Aug 06. After the screening visit, the patients that met inclusion and exclusion criteria were selected to participate in the study. The last patient out was in Jul 07.
Pre-assignment Details: A wash out period was needed in case of a previous inefficient antihypertensive medication, so it was interrupted from 2 to 3 wks before the enrollment. The patient could be excluded considering the exclusion criteria.
Groups:
- Olmesartan + Hydrochlorothiazide + Amlodipine: 1. olmesartan monotherapy was the starting dosage regimen. Blood pressure (BP) measurments were obtained at 4, 8 and 9 weeks. If BP goals were not met at a measurment point the participant's medication was elevated to the next step and BP measurments taken at the next 4, 8, and 9 weeks.
  2. olmesartan 20 mg/ hydrochlorothiazide 12.5 mg tablets was the first titration regimen if blood pressure goals were not achieved
  3. olmesartan 40 mg + hydrochlorothiazide 25 mg tablets was the second titration regimen if blood pressure goals were not achieved
  4. olmesartan 40 mg + hydrochlorothiazide 25 mg tablets + amlodipine 5 mg tablets was the third titration regimen if blood pressure goals were not achieved
Period: Overall Study
Arm/Group | Olmesartan + Hydrochlorothiazide + Amlodipine
Started | 144
Completed | 124
Not Completed | 20
Not completed — Lack of Efficacy | 20

BASELINE CHARACTERISTICS:
Arm/Group | Olmesartan + Hydrochlorothiazide + Amlodipine
Number analyzed (Participants) | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 132
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 70
Race/Ethnicity, Customized [Number; unit: Participants]
  Black | 24
  White | 83
  Asian | 7
  Other | 30
Region of Enrollment [Number; unit: participants]
  Brazil | 144

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Achieved a Blood Pressure Goal of Less Than 130/85 (Olmesartan 20 mg Monotherapy)
Description: Number of patients that achieved a blood pressure (BP) goal of less than 130/85 in the first group (olmesartan monotherapy 20 mg). If BP was > or = to 140/90 at 4,8, or 9 wks the participant went to next level for an additional 4-9 weeks at the next medication level
Time Frame: 4 - 9 wks of olmesartan monotherapy
Population: In this first dosage group 144 started and 38 patients met their blood pressure goal; therefore, 106 started the first titration regimen. There were no dropouts.
Measure: Number; unit: Participants
Groups:
- Olmesartan Monotherapy: olmesartan monotherapy 20 mg for 4-9 weeks based on blood pressure (BP) measurements at 4, 8 or 9 weeks. Participant went to next treatment if BP > or = to 140/90 mm Hg
Arm/Group | Olmesartan Monotherapy
Number analyzed (Participants) | 144
Participants | 38

2. Primary Outcome: Number of Patients That Achieved a Blood Pressure Goal of Less Than 130/85 in First Titrated Group (Olmesartan 20 mg + 12.5 mg Hydrochlorothiazide)
Description: Number of patients that achieved a blood pressure goal of less than 130/85 in first titrated group (olmesartan 20 mg + 12.5 mg hydrochlorothiazide)If BP was > or = to 140/90 at 4,8, or 9 wks the participant went to next level of medication for an additional 4-9 weeks
Time Frame: 4 to 9 weeks on combination therapy
Population: In this first titration group 106 patients started and 33 achieved their blood pressure goal. There were no dropouts and 73 subject started the second titration regimen.
Measure: Number; unit: Participants
Groups:
- Olmesartan + Hydrochlorothiazide: olmesartan 20 mg/hydrochlorothiazide 12.5 mg tablets for 4-9 weeks based on blood pressure (BP) measurements at 4, 8 or 9 weeks. Participant went to next treatment if BP > or = to 140/90 mm Hg
Arm/Group | Olmesartan + Hydrochlorothiazide
Number analyzed (Participants) | 106
Participants | 33

3. Primary Outcome: Number of Patients That Achieved a Blood Pressure Goal of Less Than 130/85 in Second Titrated Group (Olmesartan 40 mg + 25 mg Hydrochlorothiazide)
Description: Number of patients that achieved a blood pressure goal of less than 130/85 in second titrated group (olmesartan 40 mg + 25 mg hydrochlorothiazide). If BP was > or = to 140/90 at 4,8, or 9 wks the participant went to next level of medication for an additional 4-9 weeks.
Time Frame: 4 to 9 weeks
Population: 73 patients started the second titration regimen and 41 met their blood pressure goal. There were no dropouts. 32 started the final titration regimen.
Measure: Number; unit: Participants
Groups:
- Olmesartan + Hydrochlorothiazide: olmesartan 40 mg/+ hydrochlorothiazide 25 mg tablets for 4-9 weeks based on blood pressure (BP) measurements at 4, 8 or 9 weeks. Participant went to next treatment if BP > or = to 140/90 mm Hg
Arm/Group | Olmesartan + Hydrochlorothiazide
Number analyzed (Participants) | 73
Participants | 41

4. Primary Outcome: Number of Patients That Achieved a Blood Pressure Goal of Less Than 130/85 in Third Titrated Group (Olmesartan + Hydrochorothiazide + Amlodipine)
Description: Number of patients that achieved a blood pressure goal of less than 130/85 in third titrated group (olmesartan 40 mg + 25 mg hydrochlorothiazide + amlodipine 5 mg). This combination was maintained as long as the participant's blood pressure remained within predefined parameters. If not, participant discontinued for lack of efficacy.
Time Frame: 4 - 9 weeks
Population: 32 subjects started the third and final titration regimen and 12 met their blood pressure goals. 20 dropped out for lack of efficacy.
Measure: Number; unit: Participants
Groups:
- Olmesartan + Hydrochlorothiazide + Amlodipine: olmesartan 40 mg/+ hydrochlorothiazide 25 mg tablets + amlodipine tablets 5 mg for 4-9 weeks based on blood pressure (BP) measurements at 4, 8 or 9 weeks. Participant went to next treatment if BP > or = to 140/90 mm Hg
Arm/Group | Olmesartan + Hydrochlorothiazide + Amlodipine
Number analyzed (Participants) | 32
Participants | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No